CLINICAL TRIAL: NCT05890859
Title: Lean Body Mass in Head and Neck Cancer Patients During Cisplatin-based Chemoradiation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Department of Public Health, Denmark (Other)
Responsible Party: Principal Investigator, Simon Lønbro, PhD, Department of Public Health, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LBM in HNSCC during treatment
Record Dates: First submitted 2023-05-16; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Head and Neck Cancer Patients; Lean Body Mass; Body Composition Changes
Keywords: lean body mass; body composition; muscle strength; functional performance; cisplatin; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Absorptiometry, Photon; Exercise Test

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DXA scans and physical tests (Other): All patients are allocated to this arm and will undergod DXA scans and physical testing in addition to usual care/treatment
  Interventions: Diagnostic Test: DXA scan; Behavioral: Physical testing

INTERVENTIONS:
Diagnostic Test: DXA scan — The patients will undergo 5 DXA scans fro pre- to post treatment
Behavioral: Physical testing — The patients will undergo tests for maximal muscle strength and functional performance before and after treatment

SUMMARY:
The goal of this clinical trial is to investigate the changes in body composition in head and neck cancer patients during treatment. The main questions it aims to answer are: What is the rate of lean body mass loss and how is it associated with changes in muscle strength and functional performance? Is the lean body mass loss impacted by adding chemotherapy to the radiation treatment? Participants will be asked to undergo five body composition scans during treatment and undergo tests for muscle strength and functional performance before and after treatment.

DETAILED DESCRIPTION:
The primary aim of the present study is to investigate the rate of decline in body composition (LBM, body weight and fat mass) as well as changes in maximal muscle strength and functional performance during radiation treatment in HNSCC patients and to investigate the association between the loss of LBM and impairments in maximal muscle strength and functional performance. Secondly, the study investigates whether adding cisplatin during chemoradiation induces exacerbated LBM loss compared to radiation alone.

50 patients are expected to be included in the study. Inclusion criteria are: (1) histologically proven squamous cell carcinoma of the larynx, pharynx, or oral cavity, (2) prescribed to radical or post-operative radiotherapy of at least 60 Gy with or without concomitant chemotherapy. Exclusion criteria were palliative radiation or participation in competing research protocols.

Five times during treatment (biweekly), patients will be asked to undergo a Dual Energy X-ray Absorptiometry scan to evaluate changes in lean body mass and fat mass. Before and after treatment patients are asked to perform three test for maximal muscle strength (one repetition maximum knee extension, chest press and leg press) as well as three functional performance test (30 s arm curl, 30 s chair rise and stair climb).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven squamous cell carcinoma of the larynx, pharynx, or oral cavity
* Prescribed to radical or post-operative radiotherapy of at least 60 Gy with or without concomitant chemotherapy

Exclusion Criteria:

* Palliative radiation or participation in competing research protocols

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-04-05 (Actual); Primary Completion 2017-07-31 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Lean body mass | Bi-weekly from treatment start to two weeks post treatment (5 scans in total)
  Lean body mass in kg determined by DXA scans

SECONDARY OUTCOMES:
Fat mass | Bi-weekly from treatment start to two weeks post treatment (5 scans in total)
  FAt mass in kg measured by DXA scans

OTHER OUTCOMES:
Maximal muscle strength | Before and after treatment (i.e. 2-3 days before treatment start and two weeks after treatment end)
  One repetition maximum in knee extension (unilateral), leg press (unilateral) and chest press (bilateral)
Stair climb performance | Before and after treatment (i.e. 2-3 days before treatment start and two weeks after treatment end)
  The fastest walking/running time in a stair climb test is recorded (two flights of stairs)
Arm curl performance | Before and after treatment (i.e. 2-3 days before treatment start and two weeks after treatment end)
  The maximum number of repetitions in 30 s arm curl test are recorded
Chair rise performance | Before and after treatment (i.e. 2-3 days before treatment start and two weeks after treatment end)
  The maximum number of repetitions in 30 s chair rise test are recorded

CONTACTS AND LOCATIONS:
Overall Officials: Simon Lønbro, PhD, Principal Investigator — University of Aarhus
Locations (1):
- Odense University Hospital, Odense C, Southern Denmark Region, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lonbro S, Gam S, Hermann AP, Hansen CR, Johansen J. Accelerated loss of lean body mass in head and neck cancer patients during cisplatin-based chemoradiation. Acta Oncol. 2023 Nov;62(11):1403-1411. doi: 10.1080/0284186X.2023.2245558. Epub 2023 Aug 17. PMID 37589161